CLINICAL TRIAL: NCT01338636
Title: An Open-Label Uncontrolled Study of the Safety and Efficacy of Ambrisentan in Patients With Exercise Induced Pulmonary Arterial Hypertension
Brief Title: An Open-Label Uncontrolled Study of the Safety and Efficacy of Ambrisentan in Participants With Exercise-Induced Pulmonary Arterial Hypertension (PAH)
Acronym: EiPAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Aaron Waxman MD PhD, Director, Pulmonary Vascular Disease Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008P000687
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Exercise-induced Pulmonary Arterial Hypertension
Keywords: Exercise-induced pulmonary arterial hypertension (EIPAH); Pulmonary arterial hypertension (PAH); ambrisentan; Advanced cardiopulmonary exercise test (CPET)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Exercise-induced PAH (Other): Open-label ambrisentan
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — 5 mg orally every day for 4 weeks. At Week 4, if ambrisentan 5 mg was tolerated, the dose was increased to 10 mg every day for the remainder of the 24-week period.
  Other Names: Letairis

SUMMARY:
The purpose of this study is assess whether ambrisentan can help people with exercise- induced pulmonary arterial hypertension (EIPAH). The investigators also want to find out if ambrisentan is safe to take without causing excessive side effects.

DETAILED DESCRIPTION:
EIPAH population: These participants may provide a unique window into the pathogenesis of PAH. Our data suggest that these participants may represent an early phase of PAH with an abnormal vascular response.

The study includes an assessment of the potential impact of ambrisentan on the exercise capacity Advanced Level-3 cardiopulmonary exercise test (CPET) and the World Health Organization functional class (WHO FC).

ELIGIBILITY:
Inclusion Criteria:

* The participant provides written informed consent before the commencement of any study related procedure.
* The participant is 18 years of age or older.
* If a female participant of child-bearing potential, the participant must agree to use 2 forms of contraceptive therapy, including at least 1 barrier method, throughout the study and follow-up. (Women who are surgically sterile or those post-menopausal for at least 2 years are not considered to be of childbearing potential.)
* The participant has findings of either exercise induced PAH on an Advanced Level-3 CPET performed within the last 6-months and is a New York Heart Association (NYHA) Class I or II.
* The participant has a left ventricular ejection fraction (LVEF) of 55%, obtained by any appropriate method (i.e., echocardiographic assessment (ECHO), radionuclide imaging, or cardiac catheterization)
* The participant is taking a stable concomitant medication regimen for at least 4 weeks prior to enrollment in the study that is not expected to change during the study period and follow-up. Changes in diuretic and/or nitrate therapy as needed during the study period are acceptable.

Exclusion Criteria

* The participant has clinically significant psychiatric, addictive, neurologic disease or any other condition that, in the Investigator's opinion, would compromise his/her ability to give informed consent, participate fully in this study, or prevent adherence to the requirements of the study protocol.
* The participant has evidence of unstable cardiovascular disease including intermittent atrial fibrillation or unstable angina within the 4 weeks prior to Screening.
* The participant has diagnosis of exercise induced heart failure with preserved ejection fraction (previously diastolic dysfunction).
* The participant has amyloidosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis.
* The participant has a history of myocardial infarction, coronary artery bypass graft surgery, or percutaneous cardiac intervention within the last 3 months.
* The participant has clinically significant valvular heart disease in the opinion of the Investigator.
* The participant has a history of cerebrovascular accident or transient ischemic attack within the last 3 months.
* Participant has a serum alanine transaminase (ALT) or aspartate transaminase (AST) lab value that is greater than 1.5x upper limit of normal (ULN) prior to Baseline Visit.
* Participant has discontinued other endothelial receptor agonist (ERA) treatment (e.g. bosentan) for any adverse event.
* The participant has, in the opinion of the Investigator, a dependence on alcohol.
* The participant has, in the opinion of the Investigator, a dependence on illicit drugs.
* The participant has anemia defined as hemoglobin (Hgb) below 10.0 g/dL.

  * A participant may qualify for the study following diagnosis and treatment of anemia, if the anemia is due to iron and/or vitamin deficiency.
* The participant has exercise tolerance limited by noncardiac causes (e.g., exercise-induced asthma, chronic obstructive pulmonary disease, malignancy, obesity, musculoskeletal disorder).
* The participant has uncontrolled systemic hypertension defined as a resting blood pressure of 140/90 mmHg if on no treatment for systemic hypertension or 160/90 mmHg if on 2 systemic hypertension medications. For participants who are receiving treatment for diabetes mellitus, uncontrolled systemic hypertension is defined as ≥ 130/80 mmHg.
* The participant has the presence, or history, of malignancy that required significant medical intervention within the preceding 3 months and/or is likely to result in death within the next 2 years.
* The participant has chronic renal impairment or renal insufficiency defined by a serum creatinine 2.5 mg/dL and/or the requirement for dialysis.
* The participant is lactating, breastfeeding, or pregnant.
* The participant received any chronic prostacyclin, prostacyclin analogue, ERA, or phosphodiesterase (PDE) inhibitor therapy within the 30 days prior to study entry. The use of PDE inhibitors "as needed" for erectile dysfunction is acceptable as long as the participant is not dosed within 24 hours of an efficacy assessment.
* The participant has a documented allergy to Lidocaine.
* Have received any investigational medication within 30 days prior to the start of this study or be scheduled to receive another investigational drug during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Waxman, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise-induced PAH: Ambrisentan 5 mg orally every day for 4 weeks. At Week 4, if ambrisentan 5 mg was tolerated, the dose was increased to 10 mg every day for the remainder of the 24-week period.
Period: Overall Study
Arm/Group | Exercise-induced PAH
Started | 30
Completed | 22
Not Completed | 8
Not completed — Withdrawn due to lack of improvement | 8

BASELINE CHARACTERISTICS:
Population: The analysis population included all participants.
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.12 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Peak Exercise Mean Pulmonary Artery Pressure (mPAP), Transpulmonary Pressure Gradient (TPG), and Pulmonary Capillary Wedge Pressure (PCWP)
Description: mPAP is measure of the blood pressure found in the main artery of the lung. TPG is the difference between mean pulmonary arterial pressure and left atrial pressure. PCWP is the pressure measured by wedging a pulmonary catheter with an inflated balloon into a small pulmonary arterial branch.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
mmHg
  mPAP | -5.2 (5.6)
  TPG | -7.1 (8.0)
  PCWP | 2.9 (5.6)

2. Primary Outcome: Change From Baseline in Peak Exercise Pulmonary Vascular Resistance (PVR)
Description: PVR is the resistance offered by the pulmonary circulatory system.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: Woods units (WU)
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
Woods units (WU) | -0.9 (0.7)

3. Primary Outcome: Change From Baseline in Peak Exercise Pulmonary Vascular Compliance (PVC )
Description: PVC is a measure of a pulmonary vein's ability to expand.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: mL/mmHg
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
mL/mmHg | 0.8 (1.4)

4. Primary Outcome: Change From Baseline in Peak Exercise Cardiac Output (CO)
Description: CO is the amount of blood pumped by the heart per minute.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
L/min | 2.3 (1.4)

5. Primary Outcome: Change From Baseline in Peak Exercise Maximum Oxygen Uptake (VO2max)
Description: VO2max is the measurement of the maximum amount of oxygen that an individual can utilize during intense or maximal exercise.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
percent predicted | 4.4 (2.6)

6. Secondary Outcome: Change From Baseline in 6-minute Walk Distance (6MWD)
Description: 6MWD is the distance walked by the participant in 6 minutes.
Time Frame: Baseline to Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
meters | 34.8 (73.2)

7. Secondary Outcome: Borg Dyspnea Scale Score
Description: The Borg Dyspnea Scale measures how breathless the participant feels. Scores range from 0 (no shortness of breath) to 10 (more short of breath than ever experienced). (minimum score 0, maximum score 10 with 10 being worsening outcome)
Time Frame: Baseline and Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
score on a scale
  Baseline | 5.1 (2.8)
  Week 24 | 3.0 (0.9)

8. Secondary Outcome: World Health Organization Functional Class (WHO FC)
Description: The WHO FC categorizes cardiac disability using four classes, ranging from Class 1 (without limitation of physical activity) to Class 4 (inability to carry on any physical activity without discomfort).
Time Frame: Baseline and Week 24
Population: The analysis population included evaluable participants who completed the 24-week treatment period.
Measure: Mean (Standard Deviation); unit: class
Arm/Group | Exercise-induced PAH
Number analyzed (Participants) | 22
class
  Baseline | 2.0 (0.6)
  Week 24 | 1.5 (0.6)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Exercise-induced PAH
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 25/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise-induced PAH (N=30)
Peripheral edema (Metabolism and nutrition disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Headache (Nervous system disorders) | 5
Flushing (Vascular disorders) | 4
Increased cough (Respiratory, thoracic and mediastinal disorders) | 4
Joint and body pain (Musculoskeletal and connective tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Gastrointestinal infection (Gastrointestinal disorders) | 2
Jaw pain (Musculoskeletal and connective tissue disorders) | 1
Nose bleed (Vascular disorders) | 1
Palpitations (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Worsening dyspnea on exertion (Cardiac disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes